CLINICAL TRIAL: NCT01515891
Title: An Open-label Study in Healthy Male Subjects to Assess the Absorption, Distribution, Metabolism and Excretion of [14C]-Labeled BIA 9-1067 and Metabolites Following a Single-dose Oral Administration
Brief Title: Absorption, Distribution, Metabolism and Excretion of [14C]-Labeled BIA 9-1067 and Metabolites
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-103
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2014-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BIA 9-1067 (Experimental): 90 µCi (3.33 MBq) [14C]-labeled of 100 mg BIA 9-1067 (single-dose).
  Interventions: Drug: BIA 9-1067

INTERVENTIONS:
Drug: BIA 9-1067 — 90 µCi (3.33 MBq) [14C]-labeled of 100 mg BIA 9-1067 (single-dose).
  Other Names: Opicapone

SUMMARY:
To determine the absorption, metabolism and excretion of BIA 9-1067.

DETAILED DESCRIPTION:
Monocentre, open, non-placebo-controlled, single-group, single-dose study

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian male subjects, 40-55 years of age.
* Sitting blood pressure and pulse rate within a clinically acceptable range for the purposes of the study, i.e.: BP: 100 - 160 mmHg systolic, 50 - 95 mmHg diastolic and pulse rate: 50 - 100 bpm. Blood pressure and pulse were to be measured after 3 minutes resting in a sitting position.
* Subject body mass index was to be between 18 and 28 kg/m2
* Normal 12-lead ECG
* Ability to communicate well with the investigator and comply with the requirements of the entire study.
* The subject had given his written informed consent to participate in the study.

Exclusion Criteria:

* History of serious adverse reactions or hypersensitivity to any drug.
* Presence or history of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis).
* History of alcohol or drug abuse in the last 5 years.
* Abnormal physical findings of clinical significance at the screening examination or baseline which would interfere with the objectives of the study.
* Need of any prescription medication within 14 days prior to the administration of the drug and/or nonprescription medication within 7 days prior to the administration of the drug.
* Participation in other clinical trials during the previous month in which an investigational drug or a commercially available drug was tested.
* Loss of 500 mL blood or more during the 3 month period before the study, e.g., as a donor.
* Existence of any surgical or medical condition which might interfere with the absorption, distribution, metabolism or excretion of the drug, i.e., impaired renal or hepatic function, diabetes mellitus, cardiovascular abnormalities, chronic symptoms of pronounced constipation or diarrhoea or conditions associated with total or partial obstruction of the urinary tract.
* Symptoms of a significant somatic or mental illness in the 4 week period preceding drug administration.
* History of hepatitis B and / or C and / or positive serology results which indicate the presence of hepatitis B and / or C.
* Positive results from the HIV serology.
* Clinically significant abnormal laboratory values (as determined by the Principal Investigator) at the screening evaluation, however, liver parameters (SGPT, SGOT) values must be within the normal range.
* Positive results of the drug screening.
* Known hypersensitivity to BIA 9-1067.
* Heavy smokers, i.e., more than 10 cigarettes per day
* Exposure to artificial ionizing radiation in the last 12 months (e.g., x-ray investigation)
* Subject who had more than 4 flights (with more than 2 hours flight time) within the last year prior to the administration of the drug.

Ages: 40 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seiberling Michael, MD, Principal Investigator — Covance
Locations (1):
- Covance Basel Research Unit AG (formerly Swiss Pharma Contract Ltd), Allschwil, Base, Switzerland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BIA 9-1067
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BIA 9-1067
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Whole blood samples for total radioactivity analysis, plasma samples for total radioactivity analysis, and plasma samples for analysis of BIA 9-1067 and its metabolites
Time Frame: 24 hours:pre-dose and 1, 1.75, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, and 264 hours post-dose
Measure: Mean (Standard Deviation); unit: ng-eq/mL
Arm/Group | BIA 9-1067
Number analyzed (Participants) | 4
ng-eq/mL | 482.98 (265.26)

2. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: as for outcome 1
Time Frame: 24 hours at the following times: pre-dose and 1, 1.75, 2.25, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 72, 120, 168, 216, and 264 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BIA 9-1067
Number analyzed (Participants) | 4
hours | 1.69 (0.75)

3. Secondary Outcome: Area Under the Plasma-concentration Time Curve Until the Last Quantifiable Sampling Point (AUC0-t)
Description: as for outcome 1
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: h⋅ng-eq/mL
Arm/Group | BIA 9-1067
Number analyzed (Participants) | 4
h⋅ng-eq/mL | 14038.27 (4823.78)

4. Secondary Outcome: Area Under the Plasma-concentration Time Curve With Extrapolation to Infinity (AUC0-∞)
Description: as for outcome 1
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: h⋅ng-eq/mL
Arm/Group | BIA 9-1067
Number analyzed (Participants) | 4
h⋅ng-eq/mL | 33441.69 (14069.06)

ADVERSE EVENTS:
Arm/Group | BIA 9-1067
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 (N=4)
Tiredness (General disorders) | 2
Headache (Nervous system disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Loose stools (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other